CLINICAL TRIAL: NCT05858034
Title: Identifying Challenges to Healthy Aging in Persons With HIV Age 50 and Older
Brief Title: Identifying Challenges to Healthy Aging in Persons With Human Immunodeficiency Virus (HIV) Age 50 and Older
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00095309; 3P30AG021332-20 (NIH); 6 H97HA46081-01-01 (Other Grant/Funding Number: Health Resources and Services Administration)
Record Dates: First submitted 2023-04-26; First posted 2023-05-15 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-03

CONDITIONS: HIV; Aging
Keywords: human immunodeficiency virus; frailty; biomarkers of aging
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Frailty

STUDY DESIGN:
Intervention Model Description: Persons with HIV age ≥50 years followed in the Atrium Health Wake Forest Baptist Health Infectious Diseases Specialty Clinic (AHWFB IDSC), The study will take place at in the outpatient clinics of Atrium Health Wake Forest Baptist Health IDSC in Winston-Salem, NC, High Point Medical Center in High Point, NC, and Lexington Memorial Hospital (Lexington, NC).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Activity Intervention (Other): Customized selection of exercise and other community and online activity options to improve activity.
  Interventions: Other: Customized activity plan
- Nutrition Intervention (Other): Development of a customized nutrition plan to address nutritional needs.
  Interventions: Other: Customized nutrition plan

INTERVENTIONS:
Other: Customized activity plan — Clients with identified challenges to successful aging (pre-frail or frail on screening) will be invited to develop an individualized activity plan to increase mobility, strength, and stamina. Plans will combine activities to improve strength (resistance training), balance (balance exercises), and stamina, and establish weekly goals. Resistance bands and pedometers will be provided. Progress will be measured by self-reported adherence to the activity plan at week 2, 4, 8, 12 and 24 (assessed by telephone at weeks 2, 4, 8 and in person at week 12 and 24). Depression questionnaire (PHQ-9), fatigue screen, exhaustion questions, and SF-12, a measure of health-related quality of life, will be administered at baseline, week 12 and 24.
  Arms: Activity Intervention
Other: Customized nutrition plan — Participants with nutritional needs will have the option of meeting with a nutritionist to develop a personalized nutritional plan with a goal of improving diet quality and optimizing caloric intake. Progress will be measured as above.
  Arms: Nutrition Intervention

SUMMARY:
The primary objective of this study is to identify and characterize frailty and pre-frailty in persons age 50 and older living with human immunodeficiency virus (HIV) followed by the Atrium Health Wake Forest Baptist Infectious Diseases Specialty Clinics (IDSC).

DETAILED DESCRIPTION:
The study will implement electronic medical record-based screening for frailty (eFI), further characterize frailty using comprehensive geriatric screening, and offer a customized activity and nutrition plan to a subset of participants. Participation in phlebotomy for research biomarkers of aging is optional. The study also seeks to validate the electronic medical record embedded electronic frailty index (eFI) for the prediction of adverse outcomes in aging persons with HIV, characterize the symptoms of pre-frailty and frailty in persons followed in the IDSC, and assess the acceptability and efficacy of a customized activity and nutrition intervention targeting frailty. The study will also correlate research biomarkers of aging with aging symptoms in a subset of participants.

ELIGIBILITY:
Inclusion Criteria:

* Person living with human immunodeficiency virus (HIV)
* Age ≥50 years
* Followed by the Atrium Health Wake Forest Baptist Infectious Diseases Specialty Clinic (IDSC)
* Eligible for Ryan White Program
* Able to provide informed consent
* Pre-frail or frail by electronic frailty index (eFI)

Exclusion Criteria:

* Age <50 years (study designed to characterize frailty in aging persons with HIV)
* Unable to complete the required assessments or questionnaires

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Physical Performance scores | Week 12
  Change in physical performance battery scores - Minimum score 0 - Maximum score 12 - Higher scores indicate better lower extremity function

SECONDARY OUTCOMES:
Quality of Life - 12-Item Short Form Health Survey (SF-12) Scores | Week 12
  Change in quality of life as measured by SF-12 - Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning
Percentage of Adherence with Plan | Week 12
  Reported adherence to activity and nutrition plan

OTHER OUTCOMES:
electronic frailty index human immunodeficiency virus (eFI-HIV) scores | Baseline
  categorized as fit (eFI ≤0.10), pre-frail (0.10 < eFI≤0.21), and frail (eFI > 0.21) - the greater the score, the increased frailty
Comprehensive geriatric screening (CGS) - Short Physical Performance Battery | Week 12
  Short performance battery score (0-12) - The SPPB total score ranges from 0 (worst performance) to 12 points (best performance) and categorically evaluates performance in the tests using three or four classes of scores: three classes: 0-6 points (poor performance), 7-9 points (moderate performance), and 10-12 points (good performance)
Comprehensive geriatric screening (CGS) - Pepper Assessment Tool for Disability (PAT-D) Scores | Week 12
  self-reported mobility, basic and instrumental activities of daily living - Responses are made on a five-point Likert scale ranging from 1 ("usually did with no difficulty") to 5 ("unable to do") or a box can be checked that reads "usually did not do for other reasons".
Comprehensive geriatric screening (CGS) - brief cognitive screen (Mini-Cog) Scores | Week 12
  (Total Possible Score: 0-5) - A total score of 0, 1, or 2 indicates higher likelihood of clinically important cognitive impairment. A total score of 3, 4, or 5 indicates lower likelihood of dementia but does not rule out some degree of cognitive impairment.
depression Patient Health Questionnaire (PHQ-9) Scores | Week 12
  Scores less than 5 almost always signified the absence of a depressive disorder; scores of 5 to 9 predominantly represented patients with either no depression or subthreshold (i.e., other) depression; scores of 10 to 14 represented a spectrum of patients; and scores of 15 or greater usually indicated major depression.
anxiety questionnaire - General Anxiety Disorder-7 (GAD-7) Scores | Week 12
  Scoring GAD-7 Anxiety Severity. This is calculated by assigning scores - GAD-7 total score for the seven items ranges from 0 to 21. 0-4: minimal anxiety.
fatigue/exhaustion survey scores | Week 12
  The fatigue/exhaustion questions will be administered using a paper survey

CONTACTS AND LOCATIONS:
Overall Officials: Caryn G Morse, MD, MPH, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months after completion of the study.
Access Criteria: Principal investigator permission and Institutional Review Board (IRB) review required.